CLINICAL TRIAL: NCT05369845
Title: Evaluation of Prognostic Criteria for Observance of Continuous Positive Pressure for the Treatment of Obstructive Sleep Apnea Syndrome
Brief Title: Observance of Continuous Positive Pressure for the Treatment of Obstructive Sleep Apnea Syndrome
Acronym: EvOPPC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2022_843_0007
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea Syndrome; Continuous Positive Airway Pressure; Adherence; Perception and Beliefs
Keywords: Obstructive Sleep Apnea Syndrome; Continuous Positive Airway Pressure; Adherence; Perception and Beliefs
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: questionary — the patient will complete validated questionnaires, at three periods (at the time of the initiation of the CPAP, and during the 2 planned follow-up consultations: four months and at 1 year) The validated questionnaires are as follows: Illness Perception Questionnaire (IPQ-R), Beliefs about Medicines Questionnaire (BMQ), Morisky Medication Adherence Scale (MMAS), Hospital Anxiety and Depression Scale (HADS), Rollnick Scale.

SUMMARY:
Moderate to severe obstructive sleep apnea syndrome (OSAS) (HAI hypopnea apnea index ≥ 15) is a common pathology, which affects 6 to 17% of the general population. The Alaska study, which involved 480,000 apneic patients newly fitted with CPAP, showed that 76.9% of patients were still under treatment for one year, 62.9% after two years, and 52.3% after three years.

All patients who recently diagnosed with OSAS in the Sleep Disorder Unit (unity de Pathologies du Sommeil et de la Vigilance, CHU d'AMIENS-PICARDIE, FRANCE) and who are requiring CPAP will be included. On the day of their hospitalization for the implementation of the CPAP therapy, patients will answer validated questionnaires to assess their level of motivation and adherence to the initiation of treatment but also to assess their knowledge and understanding of the disease and its treatment. These questionnaires will be repeated at the four-month and one-year follow-up consultations (+/- 21 days).

The aim of the study is to identify the prognostic factors of adherence to CPAP, leading to a better understanding and management of patients with sleep apnea syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old)
* Diagnosis of moderate to severe obstructive sleep apnea syndrome OSAS (AHI ≥ 15) by polygraphy or polysomnography performed in our Sleep disorder Unit
* Requiring CPAP therapy
* Informed consent

Exclusion Criteria:

* Patient previously treated with CPAP therapy
* Psychiatric illness destabilized
* Unstable medical condition (i.e. COPD exacerbation, acute cardiac dysfunction, etc.)
* Planned obesity or ENT surgery (because CPAP treatment is planned for a short period)
* Central or mixed apnea syndrome
* Patient under 18 years old
* Pregnant, parturient or breastfeeding woman
* Patient under guardianship, curators or deprived of liberty
* Patient participating in another research including an exclusion period still in progress at the pre-inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2022-05-05 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time (in minutes) for the daily use of the CPAP therapy | at 4 weeks
Time (in minutes) for the daily use of the CPAP therapy | at 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No